CLINICAL TRIAL: NCT05743946
Title: Evaluating Trikafta for the Treatment of Patients With Non-cystic Fibrosis Bronchiectasis (NCFBE)
Brief Title: Trikafta for Patients With Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, Eric Sorscher, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004736
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
MeSH Terms: interventions — elexacaftor, ivacaftor, tezacaftor drug combination; elexacaftor; tezacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trikafta (Experimental): Participants with NCFBE and one known CFTR mutation and/or mildly elevated sweat chloride measurements (i.e., 30-60 mEq/L) receiving Trikafta for four weeks.
  Interventions: Drug: Trikafta

INTERVENTIONS:
Drug: Trikafta — Participants will be given elexacaftor 100 mg/tezacaftor 50 mg/ivacaftor 75 mg (two pills once daily in the morning) and ivacaftor 150 mg (once daily in the evening), as the FDA-registered agent, Trikafta. Dose and schedule will be for 28 days, and otherwise identical to what has already been FDA-approved for effective treatment of cystic fibrosis.
  Other Names: elexacaftor; tezacaftor; ivacaftor

SUMMARY:
Study participants with non-cystic fibrosis bronchiectasis will be given Trikafta for four weeks. The researchers will monitor clinical endpoints, quality of life, and weight. Additionally, cutaneous punch biopsy material material or blood samples from participants who agree to do this optional test will be collected to test cellular response to Trikafta.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis (NCFBE) is a clinical syndrome characterized by abnormal dilatation of the airways, airflow obstruction, persistent cough, excessive sputum production and recurrent lung infections. In terms of pathophysiology, airway dilatation and other features are associated with impaired mucociliary clearance and failure to adequately expel bacteria and mucus secretions from the airways. These events contribute to persistent infection, inflammation, and further progressive airway damage, leading to diminished lung function and eventually may cause respiratory failure and death. The pathogenesis of NCFBE is complex, poorly understood, and is likely to vary depending on the underlying etiology and important modifying factors.

Trikafta is approved for patients with cystic fibrosis (CF) carrying at least one copy of the common F508del variant or a number of other cystic fibrosis transmembrane conductance regulator (CFTR) mutations. Trikafta is a combination of three CF drugs, elexacaftor, ivacaftor, and tezacaftor, that helps CFTR proteins work more effectively. Patients with common forms of CF typically exhibit a robust pulmonary benefit from Trikafta within several days to a few weeks of initiating treatment.

NCFBE is clinically and pathologically similar to certain features of cystic fibrosis lung disease. Patients with NCFBE are not approved for Trikafta, and do not have access to the drug. Based on a considerable body of evidence, the researchers believe: 1) cutaneous punch biopsy material and/or blood sample, differentiated to airway epithelium, can be used to identify patients with NCFBE likely to benefit from drugs such as Trikafta, and 2) many patients with NCFBE have a disease likely to exhibit significant clinical improvement when treated with a drug such as Trikafta that activates CFTR-dependent ion transport, although neither of those notions has been adequately tested or proposed previously.

This study is an open-label, single center trial of orally administered elexacaftor, tezacaftor and ivacaftor (Trikafta) that will enroll 30 patients with NCFBE. Study participants will have one known CFTR mutation and/or mildly elevated sweat chloride measurements. In this matter, the study will specifically and prospectively test induced pluripotent stem (iPS) cells taken from patients with NCFBE to determine in vitro thresholds for predicting CFTR rescue in vivo. Using iPS cells differentiated to exhibit a respiratory epithelial phenotype, this study will determine whether the cells can be used to predict FEV1 response among individuals with NCFBE who receive Trikafta.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Radiologic and other clinical evidence leading to a diagnosis of NCFBE
* 1 CF-causing mutation and/or sweat chloride measurement ≥ 30 mEq/L and < 60 mEq/L
* Able to perform spirometry meeting American Thoracic Society (ATS) criteria for acceptability and repeatability, and FEV1 40-90% predicted
* Clinically stable in the past 4 weeks with no evidence of bronchiectasis exacerbation
* Willingness to use at least one form of acceptable birth control including abstinence or condom with spermicide. This will include birth control for at least one month prior to screening and agreement to use such a method during study participation for an additional four weeks after the last administration of Study Drug (for postmenopausal or other women who are without the possibility of becoming pregnant, this requirement may be waived)
* Ability to take Trikafta
* Agreement to adhere to all current medical therapies as designated by the study physician

Exclusion Criteria:

* Diagnosis of cystic fibrosis
* Documented history of drug or alcohol abuse within the last year
* Pulmonary exacerbation or changes in therapy for pulmonary disease in the 4 weeks prior to screening
* Listed for lung or liver transplant at the time of screening
* Cirrhosis or elevated liver transaminases > 3 times the upper limit of normal (ULN)
* Pregnant or breastfeeding
* Inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit/grapefruit juice, or other medicines known to negatively influence Trikafta administration
* History of solid organ transplant
* Use of a cardiac pacemaker
* Active therapy for non-tuberculosis mycobacterial infection or any plan to initiate non-tuberculosis mycobacterial therapies during the study period
* Known allergy to Trikafta
* Treatment in the last 6 months with an approved CFTR modulator
* Any other condition that in the opinion of the lead investigators might confound results of the study or pose an additional risk from administering Study Drug
* Treatment with another investigational drug or other intervention within one month prior to enrollment, throughout the duration of study participation, and for an additional four weeks following final drug administration
* Evidence of cataract/lens opacity determined to be clinically significant by an ophthalmologist at or within 3 months prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Short Circuit Current Measurements in Monolayers | Baseline
  In vitro responsiveness to Trikafta is tested by determining if iPS cells that are differentiated to airway epithelia and treated with Trikafta display functional correction of CFTR expression. This is assessed by measuring short circuit currents in monolayers.
Western Blot Analysis | Baseline
  In vitro responsiveness to Trikafta is tested by determining if iPS cells that are differentiated to airway epithelia and treated with Trikafta display biological correction of CFTR expression. This is assessed by western blot analysis.
Change in Forced Expiratory Volume in One Second (FEV1) | Baseline, Day 14, Day 28, Day 56
  FEV1 provides a direct measurement of patient health and declines in FEV1 are associated with poor outcomes. FEV1 is measured by spirometry and is the maximum amount of air the participant can blow out in one second. A responder is defined as any subject with an improvement, from baseline, in FEV1 > 5% predicted. FEV1 will also be considered continuously. In this study, if at least 15% of subjects meet the definition of responder, the researchers will view this as initial evidence of a favorable result.

SECONDARY OUTCOMES:
Change in Sweat Chloride Test | Baseline, Day 14, Day 28, Day 56
  Sweat chloride concentrations of less than or equal to 29 milliequivalent per liter (mEq/L) are considered normal, while concentrations of 30-59 mEq/L are considered intermediate. Persons with CF have high levels of chloride in their sweat (concentrations ≥ 60 mEq/L mean that a diagnosis of CF is substantiated). Sweat chloride levels in persons with NCFBE are <60 mEq/L. Studying sweat chloride in persons with NCFBE will provide information regarding the effect of the study intervention using in vivo measures known to indicate CFTR rescue.
Change in Quality of Life-Bronchiectasis (QOL-B) Score | Baseline, Day 14, Day 28, Day 56
  The QOL-B is a 37-item instrument measuring symptoms and health for individuals with NCFBE. The QOL-B includes 8 scales assessing Respiratory Symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden. Responses to items are scored from 1 to 4 and scores for each scale are standardized to range from 0 to 100. A total score is not calculated. Higher scores indicate a more favorable health status.
Change in Weight | Baseline, Day 14, Day 28, Day 56
  Weight is measured in kilograms (kg).
Change in Body Mass Index (BMI) | Baseline, Day 14, Day 28, Day 56
  BMI is calculated as the body weight divided by the square of the body height measured in meters (m). BMI is expressed in units of kg/m².

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sorscher, MD, Principal Investigator — Emory University
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during this trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data will be made available for sharing immediately following publication of results from this study, with no end date.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposal should be directed to esorscher@emory.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Derived] Swenson CE, Hunt WR, Manfredi C, Beltran DJ, Hong JS, Davis BR, Suzuki S, Barilla C, Rab A, Chico C, Dangerfield J, Streby A, Barton E, Cox EM, Stecenko AA, Westbrook A, Kapolka R, Sorscher EJ. Evaluating elexacaftor/tezacaftor/ivacaftor (ETI; Trikafta) for treatment of patients with non-cystic fibrosis bronchiectasis (NCFBE): A clinical study protocol. PLoS One. 2025 Feb 14;20(2):e0316721. doi: 10.1371/journal.pone.0316721. eCollection 2025. PMID 39951444